CLINICAL TRIAL: NCT03428685
Title: A Double Blinded Randomized Controlled Trial of Early Use of Oral Progesterone in All Women for Prevention of Preterm Delivery in Singleton Pregnancy (SINPRO Study)
Brief Title: Progesterone to Prevent Preterm Delivery
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Cheung Ka Wang, Associate Consultant, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: UW 17-308
Record Dates: First submitted 2018-02-04; First posted 2018-02-12 (Actual); Last update posted 2019-04-10 (Actual); Status verified 2019-04

CONDITIONS: Preterm Birth
MeSH Terms: conditions — Premature Birth | interventions — Dydrogesterone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Active Comparator)
  Interventions: Drug: Dydrogesterone Oral Tablet
- Placebo group (Placebo Comparator)
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Dydrogesterone Oral Tablet — Oral dysdrogesteone 10mg tds will be prescribed from 12 - 36+6 weeks.
  Arms: Intervention group
Drug: Placebo Oral Tablet — Placebos will be prescribed from 12 - 36+6 weeks.
  Arms: Placebo group

SUMMARY:
Preterm birth (PTB) is a major challenge to perinatal health. It is defined as delivery before 37 completed gestational weeks. It accounts for 75% of perinatal deaths and more than 50% of long-term neurological disabilities, and it is the second most common cause of death in children under the age of 5 year. Neonates born preterm are at risk of respiratory distress syndrome, chronic lung disease, retinopathy of prematurity, necrotizing enterocolitis, intraventricular haemorrhage and sepsis in the short term, as well as cerebral palsy, motor and sensory impairment, learning difficulties, and increased risk of chronic disease in long run. It is estimated that the societal cost of PTB is $26 billion annually in the USA alone.

Until now, prevention or reduction of PTB is based on identification of risk factors in obstetrical history, biochemical markers and short cervix. History of PTB and asymptomatic short cervix at the second trimester are both strong predictors for PTB. In women with asymptomatic short cervix at the second trimester, vaginal progesterone could effectively reduce PTB. Universal cervical length screening followed by treatment with vaginal progesterone has been shown to be the most cost effective strategy in preventing PTB. These findings were confirmed in meta-analysis.

Nevertheless, only minority of women may benefit from progesterone treatment if it was being started at the second trimester. There is still a large proportion of PTB, which is currently not preventable, and the current approach to prevent PTB is far from ideal.

One possible hypothesis is that the initiation of progesterone treatment would be too late for its effect to take place. Therefore, we decide to use oral progesterone in the current study. The objective of the study is to determine whether early use of progesterone can prevent PTB better when compared with universal screening of cervical length and followed by treatment with progesterone in those with short cervix.

ELIGIBILITY:
Inclusion Criteria:

* All women age ≥ 18 years old
* Confirmed intrauterine singleton pregnancy
* Gestational age less than 14 completed weeks as defined by pelvic ultrasound

Exclusion Criteria:

* Silent miscarriage: mean gestational sac diameter ≥25 mm without fetal pole, or embryo with crown rump length ≥7 mm and no heartbeat, or no interval growth
* Suspected ectopic pregnancy
* Multiple pregnancy with silent miscarriage of one twin
* Heavy vaginal bleeding requiring surgical intervention
* Severe abdominal pain requiring surgical intervention
* Presence of fever
* History of adverse reaction to progesterone
* History of breast or genital tract malignancy
* History of suspected thromboembolic disease
* Congenital uterine anomaly
* Unwillingness or inability to comply with study procedures
* Known paternal or maternal abnormal karyotype

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1714 (Estimated)
Dates: Start 2019-01-15 (Actual); Primary Completion 2021-01 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Rate of preterm delivery | before 37+0 gestational weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Obstetrics and Gynaecology, Hong Kong, Hong Kong, China

REFERENCES:
- [Derived] Cheung KW, Seto MTY, Ng EHY. Early universal use of oral progesterone for prevention of preterm births in singleton pregnancy (SINPRO study): protocol of a multicenter, randomized, double-blind, placebo-controlled trial. Trials. 2020 Jan 30;21(1):121. doi: 10.1186/s13063-020-4067-z. PMID 32000820